CLINICAL TRIAL: NCT07131137
Title: Design and Structure of a Remote Life Balance Training Program for People With Schizophrenia
Brief Title: A Remote Life Balance Training Program for People With Schizophrenia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AtlasU
Record Dates: First submitted 2025-07-10; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Schizophenia Disorder
Keywords: schizophrenia; telerehabilitation; life balance; remote care; intervention protocol
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: The Life Balance Training Intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: The Life Balance Training Intervention — The Life Balance Training intervention is administering as an individualized, therapist-guided program over a period of eight weeks, comprising two 45-minute sessions per week conducted via videoconferencing platforms. The program's objective was to enhance engagement in meaningful daily activities, promote a sense of life balance, and improve participation in instrumental activities of daily living (IADLs). Each session focused on fundamental components, including goal setting, skills training, activity planning, and problem solving. Caregiver involvement is encouraging when appropriate to support the generalization of skills to the home environment. The sessions commenced with a collaborative goal-setting process, centred on participants' desired modifications to their daily routines and occupational balance. The curriculum encompassed a range of pertinent subjects, including meal preparation, financial management, and time management.
  Arms: Intervention group

SUMMARY:
People living with schizophrenia often experience significant disruptions to their ability to maintain a balanced lifestyle and perform daily activities. These disruptions can hinder their ability to participate successfully in community life. In response to these challenges, a pilot study was planned to examine the feasibility and effectiveness of a telerehabilitation-based occupational therapy program aimed at promoting life balance and functional skills. The eight-week intervention is delivered remotely via videoconferencing and incorporates personalized goal setting, activity planning, skills training, and problem-solving strategies tailored to each participant. Clients diagnosed with schizophrenia who could engage in virtual sessions were invited to voluntarily participate, and pre- and post-intervention assessments were planned to measure outcomes related to instrumental activities of daily living and perceived life balance. This study aims to generate preliminary data on whether a remote, therapist-guided approach can positively impact daily functioning and quality of life. This information will guide the development of larger-scale trials in the future.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of schizophrenia according to DSM-5 criteria,
* access to an Internet-enabled electronic communication device,
* a stable Internet connection.

Exclusion Criteria:

* significant communication difficulties,
* comorbid chronic neurological or psychiatric conditions,
* inability to access communication materials and the Internet.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Life Balance | 8 weeks
  Life Balance Inventory (LBI): The LBI is a self-report instrument that evaluates the congruence between the time an individual spends on 53 daily activities and the time they would prefer to spend. The assessment is comprised of two steps. First, individuals indicate whether they engage in each activity. Second, they rate their satisfaction with time spent over the past month on a 3-point scale ranging from 1 (very unbalanced) to 3 (very balanced). The LBI score, ranging from 1.00 to 3.00, is a quantitative metric that quantifies life balance. Higher scores indicate higher levels of life balance. Furthermore, four subscale scores are derived from 51 items: The scale comprises six items in the domain of health, 20 items in the domain of challenge/interest, 15 items in the domain of identity, and 10 items in the domain of relationships. The LBI demonstrates excellent internal consistency in the general population (Cronbach's α = 0.97)
Instrumental Activities of Daily Living | 8 weeks
  Lawton-Brody Instrumental Activities of Daily Living Scale (IADL): The Lawton-Brody IADL Scale is a widely used observational tool developed to assess an individual's functional competence in performing eight instrumental activities necessary for independent living. These activities include the use of the telephone, shopping, food preparation, housekeeping, laundry, transportation, medication management, and financial management. Each item is evaluated using a 3-point scale, with 1 indicating "cannot perform," 2 indicating "needs assistance," and 3 indicating "independent." The total score ranges from 8 to 24. Scores on this scale range from 8 to 24, with higher scores indicating greater independence. The scale is commonly used to make classifications, with scores of 8-10 indicating dependence, 11-16 indicating semi-dependence, and 17-24 indicating independence. The original version exhibited adequate internal consistency, as evidenced by a Cronbach's alpha of 0.85 .

CONTACTS AND LOCATIONS:
Locations (1):
- Community-based psychiatric services, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No